CLINICAL TRIAL: NCT04052698
Title: Clinical Study to Investigate the Efficacy and Safety of Wilate During Prophylaxis in Previously Treated Patients With Von Willebrand Disease (VWD)
Brief Title: Clinical Study to Investigate the Efficacy and Safety of Wilate During Prophylaxis in Previously Treated Patients With VWD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIL-31
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Von Willebrand Diseases
MeSH Terms: conditions — von Willebrand Diseases | interventions — von Willebrand Factor; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Patients with type 3, type 2 (except 2N), or severe type 1 VWD aged ≥6 years at screening receiving Wilate for prophylactic treatment.
  Interventions: Drug: Wilate

INTERVENTIONS:
Drug: Wilate — Produced from the plasma of human donors, Wilate is presented as a powder or solvent for intravenous injection containing normally 500 IU or 1000 IU human VWF and human FVIII per vial. The ratio between VWF ristocetin co-factor activity (VWF:RCo) and FVIII:C is 1:1. The product contains approximately 100 IU/ml human VWF when reconstituted with 5ml/10mL water for injection with 0.1% polysorbate 80.
  The specific activity of Wilate is ≥67 IU VWF:RCo/mg protein. The injection or infusion rate should not exceed 2-3mL per minute.
  Other Names: von Willebrand factor / Factor VIII (plasma derived)

SUMMARY:
This is a prospective, non-controlled, international, multi-center phase 3 study investigating the efficacy and safety of Wilate in previously treated adult patients with VWD, to obtain additional data on the safety and efficacy of Wilate in previously treated patients with VWD undergoing regular prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for the study:

* Aged ≥6 years at the time of screening
* VWD type 1 (baseline von Willebrand factor activity [VWF:Ristocetin Co-factor (RCo)] <30 IU/dL, 2A, 2B, 2M, or 3 according to medical history requiring substitution therapy with a VWF-containing product to control bleeding
* Currently receiving on-demand treatment with a VWF-containing product with at least 1, and an average of ≥2, documented spontaneous BEs per month in the last 6 months, with at least 2 of these BEs requiring treatment with a VWF-containing product
* Availability of records to reliably evaluate type, frequency, and treatment of BEs for at least 6 months of on-demand treatment before screening
* Female patients of child-bearing potential must have a negative urine pregnancy test at screening and agree to use adequate birth control measures; in case hormonal contra-ception is used, the medication class should remain unchanged for the duration of the study
* All patients to provide voluntarily given, fully informed written and signed consent obtained before any study-related procedures are conducted

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the study:

* Having received on-demand or prophylactic treatment with a VWF-containing product but having no records available to reliably evaluate the type, frequency, and treatment of BEs over a period of at least 6 months of on-demand treatment
* History, or current suspicion, of VWF or FVIII inhibitors
* Medical history of a thromboembolic event within 1 year before enrolment
* Severe liver or kidney diseases (alanine aminotransferase [ALAT] and aspartate trans-aminase [ASAT] levels >5 times of upper limit of normal, creatinine >120 µmol/L)
* Platelet count <100,000/µL at screening (except for VWD type 2B)
* Body weight <20 kg at screening
* Patients receiving, or scheduled to receive, immunosuppressant drugs (other than an-tiretroviral chemotherapy), such as prednisone (equivalent to >10 mg/day), or similar drugs
* Pregnant or breast-feeding at the time of enrolment
* Cervical or uterine conditions causing abnormal uterine bleeding (including infection, dysplasia)
* Treatment with any IMP in another interventional clinical study currently or within 4 weeks before enrolment
* Other coagulation disorders or bleeding disorders due to anatomical reasons
* Known hypersensitivity to any of the components of the study drug

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Solomon, Study Director — Octapharma
Locations (14):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States
- Republican Research Center for Radiation Medicine and Human Ecology, Homyel, Belarus
- Bulgaria (2):
  - "Specialized Hospital for Active Treatment of Haematological Diseases" EAD, Sofia, Sofia
  - Pediatric Clinic of Haematology and Oncology, Varna
- University Hospital Centre Zagreb, Zagreb, Croatia
- Hungary (2):
  - Medical Centre Hungarian Defence Forces, Budapest
  - Debreceni Egyetem Klinikai Központ, Regionális Haemophilia és Thrombophilia Központ, Debrecen
- Lebanon (3):
  - Hotel Dieu de France Hospital, Beirut
  - American University of Beirut Medical Center, Beirut
  - Nini Hospital, Tripoli
- Russia (2):
  - Federal State Budgetary Scientific Institution Kirov Scientific-Research Institute of Hematology and Blood Transfusion of Federal, Kirov
  - Morosovskaya Children Clinical Hospital, Moscow Health Department, Department of General Hematology with the Pathology of Hemostasis, Moscow
- Ukraine (2):
  - State Institution "National Children's Specialized Hospital "OKHMATDYT" of the Ministry of Health of Ukraine," Center of Hemostasis Pathology, Kyiv
  - Communal Nonprofit Enterprise "Western Ukrainian Specialized Children's Medical Center"of Lviv Regional Council, Lviv

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodo I, Eikenboom J, Montgomery R, Patzke J, Schneppenheim R, Di Paola J; von Willebrand factor Subcommittee of the Standardization and Scientific Committee of the International Society for Thrombosis and Haemostasis. Platelet-dependent von Willebrand factor activity. Nomenclature and methodology: communication from the SSC of the ISTH. J Thromb Haemost. 2015 Jul;13(7):1345-50. doi: 10.1111/jth.12964. Epub 2015 May 9. No abstract available. PMID 25858564
- [Background] Sadler JE. A revised classification of von Willebrand disease. For the Subcommittee on von Willebrand Factor of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Thromb Haemost. 1994 Apr;71(4):520-5. PMID 8052974
- [Background] Rodeghiero F, Castaman G, Tosetto A. How I treat von Willebrand disease. Blood. 2009 Aug 6;114(6):1158-65. doi: 10.1182/blood-2009-01-153296. Epub 2009 May 27. PMID 19474451
- [Background] Castaman G, Goodeve A, Eikenboom J; European Group on von Willebrand Disease. Principles of care for the diagnosis and treatment of von Willebrand disease. Haematologica. 2013 May;98(5):667-74. doi: 10.3324/haematol.2012.077263. PMID 23633542
- [Background] U S Department Of Health And Human Services. Opioid abuse in the United States and Department of Health and Human Services actions to address opioid-drug-related overdoses and deaths. J Pain Palliat Care Pharmacother. 2015 Jun;29(2):133-9. doi: 10.3109/15360288.2015.1037530. PMID 26095483
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Background] Maruish M. User's manual for the SF-36v2 Health Survey (3rd edition). Optum Incorporated; 2011.
- [Background] Saris-Baglama, R,DeRosa, M, Raczek, A, Bjorner, J,Turner-Bowker, D, Ware, J. The SF-10™ Health Survey for Children: A User's Guide. QualityMetric Incorporated; 2007.
- [Background] Feldman BM, Funk SM, Bergstrom BM, Zourikian N, Hilliard P, van der Net J, Engelbert R, Petrini P, van den Berg HM, Manco-Johnson MJ, Rivard GE, Abad A, Blanchette VS. Validation of a new pediatric joint scoring system from the International Hemophilia Prophylaxis Study Group: validity of the hemophilia joint health score. Arthritis Care Res (Hoboken). 2011 Feb;63(2):223-30. doi: 10.1002/acr.20353. PMID 20862683
- [Background] van Galen KPM, Timmer MA, de Kleijn P, Fischer K, Foppen W, Schutgens REG, Eikenboom J, Meijer K, Cnossen MH, Fijnvandraat K, van der Bom JG, Laros-van Gorkom BAP, Leebeek FWG, Mauser-Bunschoten EP, Win Study Group OBOT. Joint assessment in von Willebrand disease. Validation of the Haemophilia Joint Health score and Haemophilia Activities List. Thromb Haemost. 2017 Aug 1;117(8):1465-1470. doi: 10.1160/TH16-12-0967. Epub 2017 May 11. PMID 28492695
- [Background] Janssen CA, Scholten PC, Heintz AP. A simple visual assessment technique to discriminate between menorrhagia and normal menstrual blood loss. Obstet Gynecol. 1995 Jun;85(6):977-82. doi: 10.1016/0029-7844(95)00062-V. PMID 7770270
- [Background] Higham JM, O'Brien PM, Shaw RW. Assessment of menstrual blood loss using a pictorial chart. Br J Obstet Gynaecol. 1990 Aug;97(8):734-9. doi: 10.1111/j.1471-0528.1990.tb16249.x. PMID 2400752
- [Derived] Djambas Khayat C, Dubey L, Inati A, Lissitchkov T, Novik D, Peteva E, Sidonio RF Jr, Taher AT, Vilchevska KV, Vdovin V, Boban A. Efficacy and Safety of Prophylaxis With a Plasma-Derived von Willebrand Factor/Factor VIII Concentrate (Wilate) in Patients With Type 3 von Willebrand Disease-A WIL-31 Study Sub-Analysis. Eur J Haematol. 2026 Jan 30. doi: 10.1111/ejh.70117. Online ahead of print. PMID 41614378
- [Derived] Sidonio RF Jr, Boban A, Lissitchkov T, Nemes L, Vdovin V, Khayat CD. Individualizing dosing frequency may improve the efficacy of prophylaxis in patients with von Willebrand disease-a WIL-31 subanalysis. Res Pract Thromb Haemost. 2025 Oct 10;9(7):103221. doi: 10.1016/j.rpth.2025.103221. eCollection 2025 Oct. PMID 41278463
- [Derived] Sidonio RF Jr, Boban A, Dubey L, Inati A, Kiss C, Boda Z, Lissitchkov T, Nemes L, Novik D, Peteva E, Taher AT, Timofeeva MA, Vilchevska KV, Vdovin V, Werner S, Knaub S, Djambas Khayat C. von Willebrand factor/factor VIII concentrate (Wilate) prophylaxis in children and adults with von Willebrand disease. Blood Adv. 2024 Mar 26;8(6):1405-1414. doi: 10.1182/bloodadvances.2023011742. PMID 38237075
- See also: U.S Department of Health and Human Services, Health Measures — http://www.healthmeasures.net/explore-measurement-systems/promis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 43 patients were enrolled and treated at 14 study sites worldwide. Twenty-two patients had Type 3 VWD, 10 patients were aged 6-11 years, and 8 patients were aged 12-16 years. Thirty-three patients were evaluable for the primary endpoint. The sample sizes were therefore met.
Groups:
- Wilate Routine Prophylaxis in Patients With VWD: Prophylactic treatment with Wilate of previously treated patients (PTPs) with Type 3, Type 2 (except 2N), or severe Type 1 VWD.
Period: Overall Study
Arm/Group | Wilate Routine Prophylaxis in Patients With VWD
Started | 43
Safety Analysis Set (SAF) | 43 (The safety set (SAF) included all patients who received at least 1 dose of IMP.)
Modified Full Analysis Set (mFAS) | 33 (The modified full analysis set (mFAS) included all enrolled patients who received at least one dose of IMP after the baseline IVR visit in adults or the baseline PK visit in children, and excluded all patients for whom laboratory results did not confirm the patient's VWD status)
Completed | 30
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Wilate Routine Prophylaxis in Patients With VWD
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (14.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 17
  Sex: Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42
  Black or African American | 1
Height [Mean (Standard Deviation); unit: centimetres] | 161.3 (18.22)
Weight [Mean (Standard Deviation); unit: kilograms] | 62.4 (24.96)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 22.9 (6.21)
Blood Group [Count of Participants; unit: Participants]
  Blood Group A | 22
  Blood Group B | 6
  Blood Group AB | 1
  Blood Group O | 14
VWD Type [Count of Participants; unit: Participants] — Type I VWD: low levels of von Willebrand factor, and potentially lower levels of factor VIII than normal.
  Type 2 VWD: genetic mutation leading to disfunction of von Willebrand factor. Divided into subtypes 2A, 2B, 2M, and 2N, each caused by a different gene mutation.
  Type 3 VWD: low levels or no von Willebrand factor, and low levels of factor VIII.
  Participants
    Severe Type 1 VWD | 6
    Type 2 VWD | 5
    Type 3 VWD | 22
    Unconfirmed disease status | 10
No Von Willebrand Factor inhibitor history [Count of Participants; unit: Participants] | 43
No Factor VIII Inhibitor History [Count of Participants; unit: Participants] | 43
Family History of VWD [Count of Participants; unit: Participants]
  Yes | 22
  No | 21

OUTCOME MEASURES:

1. Primary Outcome: Total Annualized Bleeding Rate (TABR)
Description: The TABR was calculated as the total number of spontaneous bleeds, traumatic bleeds, and other bleeds (except menstrual bleeds) occurring in the time period between first dose of the investigational medicinal product (IMP) and the Study Completion Visit, divided by the duration (in years) between first dose of IMP and the Study Completion Visit.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: bleeding events per year
Groups:
- 6-<12 Yrs; 12-<17 Yrs; ≥17 Yrs: Age of patients
- Total: Total annualized bleeding rates in study WIL-31
Arm/Group | 6-<12 Yrs | 12-<17 Yrs | ≥17 Yrs | Total
Number analyzed (Participants) | 9 | 6 | 18 | 33
bleeding events per year | 3.73 (4.838) | 4.28 (4.647) | 6.31 (9.634) | 5.24 (7.745)

2. Primary Outcome: Comparison of Total Annualized Bleeding Rates (TABR) During Prophylaxis Treatment in Study WIL-31 to On-demand Treatment in the Same Patient Population in the Preceding Study WIL-29
Description: Estimated TABR number calculated using a negative binomial counting regression model. Comparison between this number calculated for studies WIL-29 (NCT04053699) and WIL-31. For the comparison of results from WIL-31 to WIL-29 an estimated total annualized bleeding rate was calculated for each cohort, and compared with a negative binomial counting model. As these were estimated rates, there is only one value for each cohort with no measure of spread
Time Frame: 12 Months
Measure: Number; unit: bleeding events per year
Groups:
- WIL-29 (On-demand Treatment): Includes the same patients that constitute the mFAS population in WIL-31.
- mFAS - WIL-31 (Prophylaxis Treatment): The modified full analysis set (mFAS) included all enrolled patients who received at least one dose of IMP after the baseline IVR visit in adults or the baseline PK visit in children, and excluded all patients for whom laboratory results did not confirm the patient's VWD status
Arm/Group | WIL-29 (On-demand Treatment) | mFAS - WIL-31 (Prophylaxis Treatment)
Number analyzed (Participants) | 33 | 33
bleeding events per year | 33.3751 | 5.4914
Statistical Analysis 1: Comparison: WIL-29 (On-demand Treatment) vs mFAS - WIL-31 (Prophylaxis Treatment); Test type: Non-Inferiority — 1-sided test where the mean ratio is less than 0.5 utilizing a negative binomial counting regression model. One-sided alpha level of 2.5%; p < 0.0001, Regression, Linear; Mean Difference (Final Values) = 0.1645, 95% CI 2-sided [0.10194 to 0.26558]

3. Secondary Outcome: Spontaneous Annualized Bleeding Rate (SABR)
Description: Spontaneous annualized bleeding rate (SABR) calculated in analogy with TABR
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: bleeding events per year
Groups:
- 6<12 Years; 12<17 Years; ≥17 Years: Age of participants
- Total: Total spontaneous annualized bleeding rates (SABR) across all age groups
Arm/Group | 6<12 Years | 12<17 Years | ≥17 Years | Total
Number analyzed (Participants) | 9 | 6 | 18 | 33
bleeding events per year | 2.53 (4.145) | 6 (1.49) | 4.16 (7.382) | 3.23 (5.915)

4. Secondary Outcome: Comparison of Spontaneous Annualized Bleeding Rates (SABR) During Prophylaxis Treatment in Study WIL-31 to On-demand Treatment in the Same Patient Population in the Preceding Study WIL-29.
Description: Estimated SABR number calculated using a negative binomial counting regression model. Comparison between this number calculated for studies WIL-29 (NCT04053699) and WIL-31. For the comparison of results from WIL-31 to WIL-29 an estimated total annualized bleeding rate was calculated for each cohort, and compared with a negative binomial counting model. As these were estimated rates, there is only one value for each cohort with no measure of spread
Time Frame: 12 Months
Measure: Number; unit: bleeding events per year
Arm/Group | WIL-29 (On-demand Treatment) | mFAS - WIL-31 (Prophylaxis Treatment)
Number analyzed (Participants) | 33 | 33
bleeding events per year | 24.4168 | 3.3925
Statistical Analysis 1: Comparison: WIL-29 (On-demand Treatment) vs mFAS - WIL-31 (Prophylaxis Treatment); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Regression, Linear; Mean Difference (Final Values) = 0.1389, 95% CI 2-sided [0.07664 to 0.25187]

5. Secondary Outcome: Wilate Consumption for Prophylaxis (mFAS Population)
Description: Data on the consumption of Wilate (VWF/FVIII IU/kg per month and per week per patient) for prophylactic treatment
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: IU/kilogram
Groups:
- mFAS: The modified full analysis set (mFAS) included all enrolled patients who received at least one dose of IMP after the baseline IVR visit in adults or the baseline PK visit in children, and excluded all patients for whom laboratory results did not confirm the patient's VWD status
Arm/Group | mFAS
Number analyzed (Participants) | 33
IU/kilogram
  Dose per exposure day | 31.06 (6.589)
  Dose per injection | 31.04 (6.559)
  Dose per Week in Study | 66.06 (23.359)
  Dose per Month in Study | 287.26 (101.569)

6. Secondary Outcome: Incremental In Vivo Recovery (IVR) of Von Willebrand Factor Activity (VWF:RCo)
Description: Incremental VWF:RCo IVR of Wilate over time (at baseline and at 1, 2, 3, 6, 9, and 12 months of treatment)
Time Frame: From baseline and 12-month visit
Measure: Mean (Standard Deviation); unit: kg/dL
Groups:
- mFAS Population: The modified full analysis set (mFAS) included all enrolled patients who received at least one dose of IMP after the baseline IVR visit in adults or the baseline PK visit in children, and excluded all patients for whom laboratory results did not confirm the patient's VWD status
Arm/Group | mFAS Population
Number analyzed (Participants) | 33
kg/dL
  Baseline | 1.439 (0.5259)
  12-Month Visit | 1.273 (0.6040)

7. Secondary Outcome: Incremental In Vivo Recovery (IVR) of FVIII
Description: FVIII:C of Wilate in pediatric patients (at baseline PK visit) measured by chromogenic assay
Time Frame: Baseline and 12-month visit
Measure: Mean (95% Confidence Interval); unit: kg/dL
Arm/Group | mFAS Population
Number analyzed (Participants) | 33
kg/dL
  Baseline | 1.697 [1.47 to 1.95]
  12-month visit | 2.140 [2.04 to 2.48]

8. Secondary Outcome: Efficacy of Wilate in the Treatment of Breakthrough Bleeding Events (BEs)
Description: Treatment efficacy will be assessed at the end of a BE by the patient using predefined criteria of 'Excellent', 'Good', 'Moderate' or 'None'. All effectiveness ratings assessed as either "excellent" or "good" will be considered "successfully treated".
Time Frame: 12 months
Measure: Number; unit: bleeding episodes treated
Units Other Than Participants: Bleeding events treated
Groups:
- Efficacy Assessment of Treatment of Bleeding Episodes: The efficacy assessment of bleeding episodes at the end of a BE was evaluated on a 4-point scale by the patient/legal guardian (together with the investigator in case of on-site treatment).
Arm/Group | Efficacy Assessment of Treatment of Bleeding Episodes
Number analyzed (Participants) | 33
Number analyzed (Bleeding events treated) | 121
bleeding episodes treated
  Excellent | 109
  Good | 11
  Moderate | 1
  None | 0

9. Secondary Outcome: Wilate Exposure for Prophylaxis (mFAS Population)
Description: Data on the exposure days of Wilate prophylactic treatment
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | mFAS
Number analyzed (Participants) | 33
days | 105.55 (32.782)

10. Other Pre Specified Outcome: Efficacy Rating for Wilate in Surgical Prophylaxis
Description: Efficacy will be assessed by the surgeon at the end of surgery and by the hematologist at the end of the postoperative period using predefined criteria of 'Excellent', 'Good', 'Moderate' or 'None'. In addition, an overall assessment using the 'Excellent', 'Good', 'Moderate' or 'None' scale taking both the intra- and postoperative assessments into account will be made at the end of the postoperative period by the investigator based on an algorithm.
Time Frame: 12 months
Population: A total of 3 patients had 13 surgeries that were included in the SURG population.10 of these surgeries were minor and 3 were major.
Measure: Number; unit: surgeries
Units Other Than Participants: Number of surgeries
Groups:
- Number of Surgeries: Total number of surgeries performed
Arm/Group | Number of Surgeries
Number analyzed (Participants) | 3
Number analyzed (Number of surgeries) | 13
surgeries
  Efficacy Assessment Rated 'Excellent' | 13
  Efficacy Assessment Rated 'Good' | 0
  Efficacy Assessment Rated 'Moderate' | 0
  Efficacy Assessment Rated 'None' | 0

11. Other Pre Specified Outcome: Quality of Life (QoL) Assessed Using the Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: QoL assessment based on the results from the PROMIS-29 (Patient-Reported Outcomes Measurement Information System) survey, which monitors and evaluates the physical, mental, and social health in all patients. The survey covers seven domains from the most relevant areas of self-reported health (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance and ability to participate in social roles and activities) for the majority of people with chronic illness, each domain using a scale of a minimum score of 0 and a maximum score of 10. Derived T-score values are presented with higher scores equalling higher levels of the outcome being measured (e.g. more fatigue, more physical function). T-scores were calculated using the scoring service from the HealthMeasures Assessment Center. For this T-score metric 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
Time Frame: 12 months
Population: Analysis provided on a total number of 31 completed PROMIS-29 questionnaires.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- PROMIS 29 T-Scores: For PROMIS measures, higher scores equal more of the concept being measured (e.g., more Fatigue, more Physical Function). Thus, a score of 60 is one standard deviation above the average referenced population
- Changes From Baseline: PROMIS-29 T-Scores values taken from baseline measure during participant screening
Arm/Group | PROMIS 29 T-Scores | Changes From Baseline
Number analyzed (Participants) | 31 | 31
T-score
  Physical Function | 47.63 (8.892) | 0.59 (5.457)
  Anxiety/Fear | 49.64 (7.521) | -1.47 (8.386)
  Depression/Sadness | 46.97 (7.427) | -2.15 (6.103)
  Fatigue | 47.32 (9.408) | -2.15 (8.658)
  Sleep Disturbances | 45.35 (9.884) | -1.21 (12.494)
  Ability to Participate in Social Roles/Activites | 54.20 (9.310) | 0.97 (8.472)
  Pain Interference | 51.04 (8.990) | -3.65 (7.182)

12. Other Pre Specified Outcome: Quality of Life (QoL) Assessed Using a 36-Item Short Form Health Survey, Version 2 (SF-36v2)
Description: QoL assessment based on the results from the SF-36v2 (Short Form Health Survey) questionnaire to measure functional health and well-being in patients ≥16 years. SF-36v2 ranks 8 different domains using a scale standardized with a scoring algorithm to obtain a score ranging from 0 to 100. The eight health domains include physical functioning (PF), role physical (RP), bodily pain (BP), general health problems (GH), vitality (VT), social functioning (SF), role emotional (RE) and general mental health (MH). Norm-based scoring is used for the SF-36, setting the general population mean to 50 and the SD to 10 for all scales. Scores typically range from 20 to 60, with higher scores indicating better health.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: component scores
Groups:
- Derived SF-36 Scores: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. To aid interpretation, norm-based scoring has been introduced for the SF-36, setting the general population mean to 50 and the SD to 10 for all scales.
- Changes From Baseline: SF-36 values taken from baseline measure during participant screening.
Arm/Group | Derived SF-36 Scores | Changes From Baseline
Number analyzed (Participants) | 18 | 18
component scores
  Physical Component Scores | 46.11 (10.572) | 3.58 (6.971)
  Mental Component Scores | 50.08 (10.434) | 3.82 (9.887)

13. Other Pre Specified Outcome: Quality of Life (QoL) Assessed Using a 10-Item Short Form Health Survey (SF-10)
Description: QoL assessment based on the results from a SF-10 parent-completed questionnaire for patients ≥6 and <16 years of age, in order to score physical and psychosocial health. Norm-based scoring is used for the SF-36, setting the general population mean to 50 and the SD to 10 for all scales. Scores typically range from 20 to 60, with higher scores indicating better health.
Time Frame: 12 months
Population: Analysis based on number of completed SF-10 questionnaires completed for 6-15 year old children.
Measure: Mean (Standard Deviation); unit: derived scores
Groups:
- SF-10 Scores: The SF-10 is a 10-item, parent-completed health survey for children. Higher scores indicate better health
- Changes From Baseline: SF-10 values taken from baseline measure during participant screening
Arm/Group | SF-10 Scores | Changes From Baseline
Number analyzed (Participants) | 13 | 13
derived scores
  Physical Summary Score | 40.59 (10.907) | 6.06 (13.141)
  Psychosocial Summary Score | 50.15 (7.161) | -0.48 (10.735)

14. Other Pre Specified Outcome: Joint Health Status Assessed Using Hemophilia Joint Health Score (HJHS)
Description: Joint health status will be assessed using the Hemophilia Joint Health Score (HJHS), which has been specifically validated for the assessment of the clinical outcome in VWD. HJHS evaluates six index joints to produce a score between 0-124. The maximum score for an individual index joint is 20. Higher scores indicate worse joint health.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: HJHS score
Groups:
- 6<12 Years; 12<17 Years; ≥17 Years; Total: Age of patients
Arm/Group | 6<12 Years | 12<17 Years | ≥17 Years | Total
Number analyzed (Participants) | 9 | 6 | 18 | 33
HJHS score
  Total Score (Baseline) | 0.44 (0.882) | 2.83 (5.231) | 11.47 (19.622) | 6.75 (15.168)
  Total Score (12-month) | 0.67 (2.000) | 2.67 (4.546) | 8.33 (20.780) | 4.90 (15.027)
  Total Score (Change from Baseline) | 0.22 (1.563) | -0.17 (0.983) | -4.33 (7.247) | -2.13 (5.588)

15. Other Pre Specified Outcome: Menstrual Bleeding Assessed Using Pictorial Blood Loss Assessment Chart (PBAC) Score
Description: Bleeding information from each menstrual period while in this study will be collected using the Pictorial Blood Loss Assessment Chart (PBAC). The PBAC will be provided to all female patients of child-bearing potential. The data documented in the PBAC and the investigator-calculated final score will be recorded in the electronic case report form (eCRF). The PBAC score is from 0 onwards, with no theoretical maximum. A score of >100 defines abnormal coagulation and heavy menstrual bleeding (>80ml of blood loss per menstrual cycle).
Time Frame: 12 months
Measure: Median (Standard Deviation); unit: PBAC score
Arm/Group | WIL-29 (On-demand Treatment) | mFAS - WIL-31 (Prophylaxis Treatment)
Number analyzed (Participants) | 4 | 4
PBAC score | 219.0 (91.71) | 143.5 (59.91)

ADVERSE EVENTS:
Time Frame: From patient enrolment to study completion [approximately 12 months]
Groups:
- Wilate: All patients who participated in the study and received at least 1 dose of Wilate were included in the analysis of adverse events
Arm/Group | Wilate
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 4/43
Other Adverse Events (participants affected / at risk) | 26/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Wilate (N=43)
Menorrhagia (Reproductive system and breast disorders) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Food poisoning (Gastrointestinal disorders) | 1
Haemorrhodial haemorrhage (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Wilate (N=43)
COVID-19 infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 5
Hypersensitivity (Immune system disorders) | 2
Headache (Nervous system disorders) | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Pruitus (Skin and subcutaneous tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pyrexia (General disorders) | 2
Parvovirus B19 test positive (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04052698/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04052698/SAP_001.pdf